CLINICAL TRIAL: NCT06508398
Title: Species Spectrum and Biological Properties of Bacterial and Fungal Causative Agents of Health-care-associated Infections and in Vitro Study of Antimicrobial Activity Against Them Using 4-thiazolidinone Derivatives.
Brief Title: Healthcare-Associated Infections in Ukraine and the Activity of 4-Thiazolidinone Derivatives Against Related Pathogens
Acronym: HAIsUA
Status: Completed | Type: Observational
Sponsor: Danylo Halytsky Lviv National Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 06/25/2018, N6; 06/22/2020, N6; 2020.02/0035 (Other Grant/Funding Number: National Research Foundation of Ukraine); FEMS-GO-2020-195 (Other Grant/Funding Number: Federation of European Microbiological Societies); Ministry of Health of Ukraine (Other Grant/Funding Number: 0118U000111); Ministry of Health of Ukraine (Other Grant/Funding Number: 0121U100690)
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Nosocomial Infection
Keywords: Healthcare-Associated Infections; HAIs; nosocomial infections; antimicrobial resistance; AMR; nosocomial; antibiotic resistance; device-associated pathogens; antimicrobial activity; antifungal activity; 4-thiazolidinones; thiazoles; cellular immunity; immunotropic action; guinea pigs; MALDI; rare pathogens
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — The specific types of samples that will be retained include:
  * Blood Samples: Venous blood for microbiological and biochemical analysis.
  * Urine Samples: From the urinary bladder for pathogen detection.
  * Sputum Samples: Respiratory tract microbiological testing.
  * Bronchoalveolar Lavage (BAL) Samples: From lungs to identify respiratory pathogens.
  * Wound Swabs: From wound sites for bacterial identification.
  * Oropharyngeal/Nasopharyngeal Swabs: Throat and nasal passages for pathogen detection.
  * Stool Samples: Gastrointestinal pathogen analysis. All samples will be preserved and may be used for DNA extraction to study genetic aspects of pathogen resistance and infection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patients with Healthcare-Associated Infections: This group consists of patients admitted to the Intensive Care Units (ICUs) in Lviv hospitals who are diagnosed with healthcare-associated infections (HAIs). The study involves collecting clinical samples, including blood, urine, sputum, bronchoalveolar lavage, wound swabs, and oropharyngeal/nasopharyngeal swabs, to identify bacterial and fungal pathogens and analyze their antimicrobial resistance profiles. The data collected will be used to evaluate the effectiveness of new 4-thiazolidinone derivatives against these pathogens.
  Interventions: Diagnostic Test: Microbiological Diagnostic Testing

INTERVENTIONS:
Diagnostic Test: Microbiological Diagnostic Testing — This study involves microbiological diagnostic testing of clinical samples collected from ICU patients diagnosed with healthcare-associated infections (HAIs). The intervention includes:
  Sample Collection: Blood, urine, sputum, bronchoalveolar lavage, wound swabs, and oropharyngeal/nasopharyngeal swabs.
  Pathogen Identification: Using biochemical tests, MALDI-TOF mass spectrometry, and 16S rRNA sequencing to identify bacterial and fungal pathogens.
  Antimicrobial Susceptibility Testing: Determining the resistance profiles of the identified pathogens to various antimicrobial agents.
  Evaluation of New Compounds: Testing the antimicrobial efficacy of new 4-thiazolidinone derivatives against isolated pathogens.
  This comprehensive approach aims to enhance the understanding of pathogen distribution and resistance patterns in HAIs.
  Other Names: Pathogen Identification and Antimicrobial Susceptibility Testing

SUMMARY:
The goal of this observational study is to evaluate the species spectrum and biological properties of bacterial and fungal pathogens causing healthcare-associated infections (HAIs) and to investigate the antimicrobial activity of new 4-thiazolidinone derivatives. The main questions it aims to answer are:

What are the common pathogens responsible for HAIs in ICU patients? What is the antimicrobial and antifungal efficacy of 4-thiazolidinone derivatives against these pathogens?

Participants will have their clinical samples collected and analyzed for pathogen identification and susceptibility testing. The study will involve:

Collecting clinical data and samples from ICU patients Conducting microbiological and biochemical tests Screening new antimicrobial compounds for efficacy The study does not involve a comparison group as it focuses on observational data and laboratory analysis.

DETAILED DESCRIPTION:
The study aims to characterize the structure and distribution of Healthcare-Associated Infections (HAIs) in Ukraine in recent years, features of the species spectrum of pathogens, and the spreading of antibiotic resistance, clinical and microbiological characteristics of HAIs, including those caused by rare pathogens of HAIs, as well as a search, synthesis, screening of new chemical compounds with antimicrobial and antifungal activity in order to introduce new prototypes of antimicrobial drugs.

According to the study design, and analysis of the data of the CDC of Ukraine on the registration of HAIs cases in Ukraine during 2009-2020 was conducted. As a result, for the first time in Ukraine, the registration of HAIs for the last 12 years was analyzed; according to the results, an average of 4,759 ± 710 cases of HAIs have been registered annually. The analyzed materials give grounds to claim a significant underestimation of the incidence of HAIs in the country.

According to the results of a comprehensive, dynamic, clinical, and laboratory-instrumental examination of 250 patients of 4 local hospitals' ICU departments, and based on microbiological and epidemiological criteria, the corresponding diagnosis was confirmed in 205 patients. Among persons with HAIs, 46.8% were men, and 53.2% were women. Among all cases of HAIs, 24.9% were children (including 8.8% newborns), 64.9% - people aged 18-60 years, older adults (> 60 years) were 10.2%. The most common nosologies were respiratory tract infections (36.6%) and urinary tract infections (34.1%). Most HAIs (58.6%) occurred from the 5th to the 14th day of hospital stay.

Three hundred eighty-nine biomaterials were taken, from which 309 strains of microorganisms were isolated, among which Gram-negative bacteria prevailed (51.5%), the species spectrum of which included representatives of 27 different species. Representatives of the genus Pseudomonas were the most isolated - 50 isolates, 16.2% of the total number of pathogens. Gram-positive microbiota is represented by 15 different species of pathogens, the most - members of the genus Staphylococcus - 52 isolates, which is 16.8% of the total number of pathogens. Among the fungi, 12 different species of pathogens were isolated, most of them Candida non-albicans - 20 isolates, which is 6.5% of the total number of pathogens.

For the first time in Ukraine, clinical cases caused by rare pathogens Raoultella (Klebsiella) terrigena and Vibrio metchikovii have been identified and described. Our reported cases were compared with the clinical cases described in the literature. It was shown that the isolate of R. terrigena has film-forming properties, more pronounced than the standard strain Raoutella terrigena ATCC 33257, and the rate of film formation exceeds the rate of film formation by staphylococci.

Analyzing the clinical case caused by Vibrio metchikovii, it should be noted that the most likely cause of infection is intraoperative microbial contamination of vascular prostheses.

Species identification of pathogens was performed using biochemical test systems (MIKRO-LA-TEST ErbaLachema, Czech Republic), using MALDI-TOF (conducted at the Department of Microbiology of the College of Medicine in Bydgoszcz, Poland) and for individual strains - 16sRNA-ID. The Identification score (index) of biochemical identification of cultures was > = 95%, or > = 99% for 87.4% of isolates (n=270). 50.8% of strains (n=157) had an atypicality index (Tin) of 0.25-0.49, i.e., these strains can be characterized as atypical. MALDI ID-score 95.5% of isolates (n=295) was > = 2.0, ie showed good species identification, other isolates had ID score 1.7-1.9, which indicates generic identification. PCA analysis of Gram-negative rods of the genus Klebsiella allowed to divide them into 4 main clusters and showed significant similarity of isolates and, together with RAPD analysis, allowed to confirm the in-hospital transmission of pathogens. According to the results of 16S rRNA analysis, comparisons of Klebsiella pneumoniae isolates were performed, which testified to the common origin of the infection. Different identification methods established that a complete coincidence of results were recorded for 76.1% of strains (n=235). The highest identification accuracy is shown for 16sRNA analysis, but the speed is for MALDI-TOF.

The results of the antibiotic sensitivity showed that 62.8% (n=194) of isolates were MDR, 7.4% (n=23) were EDR, 28.8% (n=89) were not-MDR. 1% (n=3) strains were attributed to PDR: 2 - P.putida and 1 - P.aeruginosa. 33.8% (n=25) of the studied enterobacteria produced ESBL from another group of 47 studied isolates (83.9%) produced OXA-48, among which all isolates were MDR. The vast majority of fungal strains (82.9%) were resistant to fluconazole, which the most common choice of this drug can explain as empirical treatment of fungal infection.

Cultures of Achromobacter xylosoxidans (№ LMU-147) and Serratia marcescens (№ LMU-48) were isolated, for which their role in causing HAIs was proved. The isolated strains are classified as class IV pathogenicity, based on UA classification (US CDC classification - Biosafety level 1), but they can penetrate internal organs, more pronounced for serration. Candida utilis (LMU-127) is a low pathogenic strain that does not have invasive properties.

Fifty-five new synthesized thiazole derivatives were used to search for and study new chemical compounds with antibiotic activity. There was a pronounced antifungal effect in 3-[5-(1H-Indol-3-ylmethylene)-4-oxo-2-thioxothiazolidin-3-yl]-propanoic acid with a minimum inhibitory concentration against fungi of the genus Candida 25 μg/mL and a selective antimicrobial effect against Escherichia coli in 2-[5-(1H-Indol-3-ylmethylene)-4-oxo-2-thioxothiazolidin-3-yl]-ethanesulfonic acid with a similar effect (MIC=25 μg/mL). The most active against Staphylococcus aureus group was 2-(5-ylidene-4-oxo-2-thioxo-thiazolidin-3-yl)-succinimides with a terminal fragment in the C5 position.

For a 2-cyano-2- [5- (ethoxymethylene) -4-oxo-3-phenyl-thiazolidin-2-ylidene] -N- (o-tolyl) acetamide derivative which does not contain a phenyleneamine or benzylidene moiety in the structure at position C5 position of the thiazolidone nucleus showed the highest activity against the multidrug-resistant clinical strain of Pseudomonas aeruginosa.

A laboratory animal model studied the immunotoxic/allergenic/acute toxic effect of the "leader compound" with antimicrobial activity. No immunotoxic and allergenic effects were found, but there is a moderate anti-inflammatory effect. Against the background of an increase in the absolute number of CD3 T-lymphocytes by 21.46%, a slight decrease in the quantitative level of CD22 B-lymphocytes (by 1.98%) was recorded. Activation of the suppressor link caused some decrease in the immunoregulatory index (indicator is unreliable).

The effect of the test substance on the level of immunoglobulins and interleukins of laboratory animals showed a significant decrease in IgA by 21.4% (p <0.05) and an increase in IgG by 21.2%. Thus, there was an increase in the activity of the phagocytic system in terms of the growth of the phagocytic number and absorption properties of neutrophils. The selectivity of such biological activity may be useful in the treatment of some immunopathological conditions.

The identified effects accompanying antifungal activity indicate the prospects for further study of the "drug-like molecule" with polytargetative action.

The analysis of the HAIs prevalence, their registration, the state of specific diagnostics, comparison of modern methods of identification of microbial isolates from clinical material indicates the need to increase the level of microbiological research, implementation of a standardized registration system, and research of nosocomial infections with potentially adverse health effects.

According to the thesis results and research of isolates' biological properties, the corresponding strains were deposited in the Depository of the Institute of Microbiology and Virology of the National Academy of Sciences of Ukraine.

Based on the research, 2 utility model patents were issued. In addition, molecular docking studies have shown that the "leader compound" 7-(3,4-Dimethoxyphenyl)-5-methyl-3H-thiazolo[4,5-b]pyridin-2-one has shown good binding to selected protein targets compared to the reference N21 inhibitor and ciprofloxacin.

Keywords Healthcare-Associated Infections (HAIs), nosocomial infections, antimicrobial resistance, antibiotic resistance, device-associated pathogens, antimicrobial activity, antifungal activity, 4-thiazolidinones, thiazoles, cellular immunity, immunotropic action, guinea pigs, MALDI, rare pathogens.

Publications. According to the thesis materials, 10 articles were published, including 8 articles indexed in the journals Web of Science and/or Scopus, article in the Ukrainian professional journal, 1 article in a non-professional journal.

The work results were presented at 17 conferences, including in the form of an oral report at 3 international conferences outside Ukraine and 1 conference in Ukraine.

Based on the work results, 2 utility model patents and 3 certificates of initial deposition of the microorganism strain were published.

ELIGIBILITY:
Inclusion Criteria:

Currently hospitalized in an ICU department. Confirmed diagnosis of a nosocomial infection (healthcare-associated infection (HAI)).

Exclusion Criteria:

Community-associated pneumonia. Infectious processes that are not related to the provision of medical care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of ICU patients from Lviv hospitals, specifically the Lviv Regional Clinical Hospital, the Military Medical Clinical Center of the Western Region, Lviv Regional Children's Clinical Hospital "Ohmatdyt," and the 8th Municipal Clinical Hospital of Lviv. These participants are diagnosed with healthcare-associated infections and will provide clinical samples for pathogen identification and antimicrobial susceptibility testing. The population includes both male and female patients across various age groups, representative of the ICU admissions at these institutions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Healthcare-Associated Infections (HAIs) | 12 months
  The primary outcome measure is to determine the incidence rate of healthcare-associated infections in ICU patients. This will be achieved by collecting and analyzing clinical samples for the presence of bacterial and fungal pathogens. The effectiveness of new 4-thiazolidinone derivatives against these pathogens will also be assessed through antimicrobial susceptibility testing.

SECONDARY OUTCOMES:
Pathogen Distribution in Healthcare-Associated Infections | 12 months
  The secondary outcome measure focuses on identifying and analyzing the distribution of bacterial and fungal pathogens causing healthcare-associated infections (HAIs) in ICU patients. This involves the collection and examination of clinical samples to determine the prevalence and types of pathogens. Additionally, the study will evaluate the antimicrobial resistance profiles of these pathogens to understand the resistance patterns and effectiveness of current treatment options.

OTHER OUTCOMES:
Clinical Outcomes of ICU Patients with HAIs | 12 months
  This measure evaluates the clinical outcomes of ICU patients diagnosed with healthcare-associated infections, including length of hospital stay, mortality rates, and readmission rates. The study aims to understand the impact of HAIs on patient recovery and hospital resource utilization.
Efficacy of 4-Thiazolidinone Derivatives | 12 months
  This measure assesses the antimicrobial and antifungal efficacy of new 4-thiazolidinone derivatives against isolated pathogens. The study involves in vitro testing to determine the minimum inhibitory concentrations (MICs) and compare them to existing treatments.
Antimicrobial Resistance Mechanisms | 12 months
  This measure investigates the genetic mechanisms of antimicrobial resistance in identified pathogens. The study involves sequencing and molecular analysis to identify resistance genes and their expression patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Yulian Konechnyi, PhD, Principal Investigator — Danylo Halytsky Lviv National Medical University
Locations (1):
- Danylo Halytsky Lviv National Medical University, Lviv, Lviv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
Access to the IPD and supporting information will be granted to researchers upon request. Researchers will need to submit a data access request form, including a brief description of their research objectives and how they intend to use the data. Data will be shared under a data use agreement to ensure proper handling and confidentiality. Researchers can request access by contacting the principal investigator via email.

REFERENCES:
- [Background] Konechnyi Y, Khorkavyi Y, Ivanchuk K, Kobza I, Sekowska A, Korniychuk O. Vibrio metschnikovii: Current state of knowledge and discussion of recently identified clinical case. Clin Case Rep. 2021 Mar 4;9(4):2236-2244. doi: 10.1002/ccr3.3999. eCollection 2021 Apr. PMID 33936672
- [Result] Lekhniuk N, Fesenko U, Pidhirnyi Y, Sekowska A, Korniychuk O, Konechnyi Y. Raoultella terrigena: Current state of knowledge, after two recently identified clinical cases in Eastern Europe. Clin Case Rep. 2021 Mar 31;9(5):e04089. doi: 10.1002/ccr3.4089. eCollection 2021 May. PMID 34026135
- [Result] Sekowska A, Konechnyi Y, Gospodarek-Komkowska E. Klebsiella pneumoniae infection in a liver transplant patient: A case report and review of the literature. Indian J Med Microbiol. 2021 Oct-Dec;39(4):548-551. doi: 10.1016/j.ijmmb.2021.07.001. Epub 2021 Jul 24. PMID 34315617
- [Result] Khamitova capital A, Cyrillic, Berillo D, Lozynskyi A, Konechnyi Y, Mural D, Georgiyants V, Lesyk R. Thiadiazole and Thiazole Derivatives as Potential Antimicrobial Agents. Mini Rev Med Chem. 2024;24(5):531-545. doi: 10.2174/1389557523666230713115947. PMID 37448365
- [Result] Konechnyi Y, Panas M, Tymchuk I, Havur O, Borysiuk O, Hubytska I, Zhurakhivska L, Konechna R, Korniychuk O. Epidemiological and microbiological aspects of healthcare-associated infections in Ukraine during the 2009-2019 period. Przegl Epidemiol. 2021;75(1):86-95. doi: 10.32394/pe.75.09. PMID 34338474
- [Result] Konechnyi Y, Rumynska T, Yushyn I, Holota S, Turkina V, Ryviuk Rydel M, Sekowska A, Salyha Y, Korniychuk O, Lesyk R. A New 4-Thiazolidinone Derivative (Les-6490) as a Gut Microbiota Modulator: Antimicrobial and Prebiotic Perspectives. Antibiotics (Basel). 2024 Mar 22;13(4):291. doi: 10.3390/antibiotics13040291. PMID 38666967